CLINICAL TRIAL: NCT02274896
Title: A Prospective Multicenter Investigation to Evaluate the Safety of the Bayston Antimicrobial Peritoneal Dialysis Catheter in ESRD Patients
Brief Title: Bayston Multicenter Antimicrobial PD Catheter Safety Study
Acronym: Bayston
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Project No Longer in Development
Sponsor: Medical Components, Inc dba MedComp (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAYPDC-14-01
Record Dates: First submitted 2014-10-17; First posted 2014-10-24 (Estimated); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: End Stage Renal Disease (ESRD)
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PD catheter group (Experimental): All patients will receive the Bayston PD catheter
  Interventions: Device: PD Catheter group

INTERVENTIONS:
Device: PD Catheter group — PD catheter

SUMMARY:
The study was designed to establish the safety of the Bayston Antimicrobial PD catheter that is impregnated with a "cocktail" of three well known anti-microbials

DETAILED DESCRIPTION:
The objective of this clinical investigation is to establish the safety of the Bayston Antimicrobial Peritoneal Dialysis Catheter in ESRD patients initiating CAPD.

The Bayston catheter is not expected to cause any safety related complications or reactions other than those described for not-impregnated peritoneal dialysis catheters. Thus the objective of this clinical investigation is to evaluate whether the Bayston catheter causes any unanticipated serious adverse device effects (USADE).

The primary hypothesis for this study is that the Bayston Antimicrobial Peritoneal Dialysis Catheter is a safe catheter for peritoneal dialysis.

No claims regarding efficacy will be verified during this clinical investigation.

This is a prospective, non-randomized, single-arm, multi-center study involving patients suffering from end stage renal disease who are eligible for treatment with peritoneal dialysis. Forty-three (43) patients will be enrolled who will be followed up to 6 months after implantation of the Bayston Antimicrobial Peritoneal Dialysis Catheter.

ELIGIBILITY:
Inclusion Criteria:

* End stage renal disease documented by clinical symptoms and/or laboratory findings
* Patients scheduled for their first PD catheter implantation
* Eligible for peritoneal dialysis (CAPD)
* Willing and able to attend all study follow-up visits
* Willing and able to understand and sign the informed consent form

Exclusion Criteria:

* A history of allergy to rifampin, trimethoprim or triclosan
* Use contact lenses or have lens implants
* Pregnant, lactating or planning to become pregnant during the course of the clinical investigation
* Recent abdominal surgery, abdominal adhesions, infected abdominal wall, diaphragmatic tears or ileus
* Respiratory insufficiency
* Infection:

  * Active infections from successful completion of antibiotic treatment for routine bacterial infection less than 4 weeks of entry into the clinical investigation (screening)
  * Febrile viral infection within 4 weeks of entry into the clinical investigation (screening)
  * Less than 12 weeks from conclusion of therapy for systemic fungal infections to screening
* Abnormal hematology parameters defined as severe anemia with hemoglobin <8.5g/dL, white blood cell count of <3,500/μl and a granulocyte count <2,000/μl
* Have collagen-vascular, connective tissue, or bleeding disorders
* Used an investigational medicinal product, biologic or device within the last 30 days prior to enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse events | 6 months
  Safety: Freedom from unanticipated serious device related adverse events up to 6 months after implantation of the Bayston catheter.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Wilkie, Dr., Principal Investigator — Renal consultant
Locations (5):
- UZ Leuven, Leuven, Belgium
- University Medical Center Utrecht, Utrecht, Netherlands
- United Kingdom (3):
  - North Bristol NHS Trust, Bristol
  - Imperial College London - Hammersmith Hospital, London
  - Sheffield Teaching Hospitals NHS Foundation Trust - Northern General Hospital, Sheffield